CLINICAL TRIAL: NCT03233438
Title: Development of a New Critical Pathway for Treatment of Acute Bacterial Skin and Skin Structure Infections
Brief Title: Development of a New Critical Pathway for Treatment of Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMO-US-ID-0528
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Bacterial Infections; Acute Bacterial Skin and Skin Structure Infection
Keywords: Critical Pathways; Health Facilities; Clinical Protocols; Patient Satisfaction; Absenteeism; Anti-Bacterial Agents; Quality of Life; Economics, Medical; Health Resources; Health resource utilization; Acute bacterial skin and skin structure infection (ABSSSI)
MeSH Terms: conditions — Bacterial Infections; Patient Satisfaction | interventions — dalbavancin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- New Critical Pathway (Active Comparator): The New Critical Pathway under study is defined as (1) use of guideline-based patient identification criteria, and, for those who meet these criteria, (2) use of dalbavancin, administered as a single intravenous (IV) dose of 1500 mg over 30 minutes for the treatment of ABSSSI.
  Interventions: Drug: Dalbavancin
- Usual Care (Active Comparator): Participants who receive Usual Care as prescribed by the physician as standard of care in clinical practice for the treatment of ABSSSI.
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin administered as a single IV dose of 1500 mg over 30 minutes.
  Other Names: Dalvance®
  Arms: New Critical Pathway
Drug: Usual Care — Usual care as prescribed by the physician as standard of care in clinical practice for the treatment of ABSSSI.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to assess the effect of a new critical pathway (use of guideline-based patient identification criteria and for those who meet these criteria, use of dalbavancin) compared to usual care for the treatment of ABSSI (Acute Bacterial Skin and Skin Structure Infections)

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients who meets the clinical definition for Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
* Known or suspected gram-positive infection.

Exclusion Criteria:

* Known or suspected gram-negative infections, anaerobic infections, or fungemia
* Known or suspected infections that are severe, life threatening or are not included in the ABSSSI Food and Drug Administration (FDA) guidance
* Injection drug users with a fever
* Severe neurological disorder leading to immobility or confined to a wheelchair
* Bilateral Lower extremity involvement of the suspected infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Gillard, Study Director — Allergan
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

REFERENCES:
- [Derived] McCarthy MW, Keyloun KR, Gillard P, Choi JJ, Pickell N, Copp R, Walsh TJ. Dalbavancin Reduces Hospital Stay and Improves Productivity for Patients with Acute Bacterial Skin and Skin Structure Infections: The ENHANCE Trial. Infect Dis Ther. 2020 Mar;9(1):53-67. doi: 10.1007/s40121-019-00275-4. Epub 2019 Nov 11. PMID 31713130
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | New Critical Pathway
Started | 48 | 43
Completed | 42 | 32
Not Completed | 6 | 11
Not completed — Lost to Follow-up | 4 | 9
Not completed — Withdrawal by Subject | 2 | 1
Not completed — No recording of dalbavancin | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population consists of all enrolled patients that has received at least one dose of antibiotics or one dose of dalbavancin for inclusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | New Critical Pathway | Total
Number analyzed (Participants) | 48 | 42 | 90
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 0 | 0 | 0
  20-29 years | 6 | 5 | 11
  30-39 years | 6 | 8 | 14
  40-49 years | 4 | 8 | 12
  50-59 years | 7 | 5 | 12
  60-69 years | 10 | 5 | 15
  70-79 years | 4 | 3 | 7
  80-89 years | 7 | 7 | 14
  90-98 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 24 | 22 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 38 | 26 | 64
  Unknown or Not Reported | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 36 | 28 | 64
  Black or African American | 1 | 7 | 8
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 0 | 0 | 0
  Patient chose not to answer | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Infection-related Total Admitted Hospital Days
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Days | 4.8 (2.55) | 3.2 (2.48)
Statistical Analysis 1: Comparison: Usual Care vs New Critical Pathway; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [0.6 to 2.6], Standard Deviation 2.5

2. Secondary Outcome: Number of Total Admitted Hospital Days
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Days | 4.9 (2.62) | 3.2 (2.48)
Statistical Analysis 1: Comparison: Usual Care vs New Critical Pathway; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [0.6 to 2.8], Standard Deviation 2.56

3. Secondary Outcome: Number of Participants With Infection-related Major Surgical Interventions That Required Operating Room Time
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  No Surgeries | 48 | 41
  Expected Surgeries | 0 | 1

4. Secondary Outcome: Number of Participants With Infection-related Hospitalizations
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  1 Occurrence | 48 | 39
  2 Occurrences | 0 | 3

5. Secondary Outcome: Number of Participants With Infection-related Hospitalizations That Resulted in Admission to Intensive Care Unit
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  Admission to ICU | 0 | 0

6. Secondary Outcome: Number of Participants With All Cause Hospitalizations in the 30 Days Post Discharge From the Hospital
Time Frame: Follow-up: 30 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  None | 47 | 39
  1 Occurrence | 1 | 3

7. Secondary Outcome: Number of Participants With Infection-related Emergency Department (ED) Visits
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  None | 46 | 40
  1 Occurrence | 2 | 2

8. Secondary Outcome: Number of Participants With Infection-related Outpatient Healthcare Visits
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  None | 26 | 20
  Any | 22 | 22

9. Secondary Outcome: Use of a Peripherally-Inserted Central Catheter (PICC) Line or Central Line to Administer Antibiotic Therapy
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  Central Line | 0 | 0
  PICC Line | 1 | 0
  Peripheral IV | 27 | 42
  No Line | 20 | 0

10. Secondary Outcome: Number of Participants With Infection-related Healthcare Visits Due to PICC Line or Central Line Used to Administer Antibiotic Therapy
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  None | 45 | 41
  1 Occurrence | 3 | 1

11. Secondary Outcome: Change From Baseline in Response to Treatment at End of Treatment Visit
Description: Response to treatment (healthcare provider assessment) comparing response at the Day 14 visit. Response to treatment will be defined through an assessment of erythema (measurement of lesion characteristics) and the absence of fever
Time Frame: Baseline, Day 14
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants
  Complete response | 24 | 24
  Partial response | 0 | 0
  Failure | 12 | 9
  Unknown | 12 | 9

12. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
Participants | 1 | 3

13. Secondary Outcome: Patient Satisfaction With Care: Overall Health
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: FAS population. 43 and 34 patients provided any survey data in the usual care group and the new critical pathway group, respectively. 40 and 32 patients completed all survey questions in the usual care group and new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
Participants
  Excellent | 2 | 8
  Very good | 16 | 10
  Good | 9 | 7
  Fair | 10 | 8
  Poor | 6 | 1

14. Secondary Outcome: Patient Satisfaction With Care: Wait in Emergency Room
Description: Patients rated their satisfaction on a 10-point scale, where 0 was the worst experience possible and 10 the best experience possible.
Time Frame: 14 Days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
scores on a scale | 5.1 (3.34) | 6.9 (3.12)

15. Secondary Outcome: Patient Satisfaction With Care: Hospitalization
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
Participants
  Yes | 43 | 34
  No | 0 | 0

16. Secondary Outcome: Patient Satisfaction With Care: Satisfaction With Hospital Stay
Description: as for outcome 14
Time Frame: 14 Days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
scores on a scale | 7.4 (2.35) | 7.4 (2.72)

17. Secondary Outcome: Patient Satisfaction With Care: Factors for Dissatisfaction With Your Hospital Stay
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: 43 & 34 patients provided any survey data in the usual care group & new critical pathway group; 40 & 32 patients completed all questions in the usual care group & new critical pathway group; 42 & 34 patients answered this question in the usual care group & new critical pathway group, respectively. Patients may have checked multiple responses.
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 42 | 34
Participants
  Hospital stay interfered with work/school | 13 | 6
  Stay got in way of daily normal activities | 17 | 8
  Stay got in the way of providing care to others | 10 | 5
  Hospital stay was expensive | 7 | 4
  Did not provide adequate monitoring by providers | 4 | 4
  Did not provide well trained healthcare providers | 3 | 1
  Hospital stay made me feel worse | 4 | 1
  Hospital stay made me feel concerned | 11 | 7
  Hospital stay was uncomfortable | 12 | 7
  Hospital stay disrupted my sleep | 24 | 10
  Other | 5 | 6
  I was not dissatisfied with my hospital stay | 12 | 12

18. Secondary Outcome: Patient Satisfaction With Care: Received IV Antibiotic Therapy for Skin Infections
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: FAS Population. 43 & 34 patients provided any survey data in the usual care group & new critical pathway group; 40 & 32 patients completed all survey questions in the usual care group & new critical pathway group; 43 & 33 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
Participants
  Yes | 43 | 33
  No | 0 | 1

19. Secondary Outcome: Patient Satisfaction With Care: Satisfaction With Receiving IV Antibiotic Therapy
Description: as for outcome 14
Time Frame: 14 Days
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 33
scores on a scale | 7.1 (2.83) | 8.1 (2.26)

20. Secondary Outcome: Patient Satisfaction With Care: Factors Contributing to Satisfaction With Receiving IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: 43 & 34 patients provided any survey data in the usual care group & new critical pathway group; 40 & 32 patients completed all questions in the usual care group & new critical pathway group; 43 & 33 patients answered this question in the usual care group & new critical pathway group, respectively. Patients may have checked multiple responses.
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 33
Participants
  Allowed me to return to work/school | 14 | 15
  Allowed me to return to daily normal activities | 15 | 20
  Allowed me to return to providing care to others | 8 | 11
  IV antibiotic therapy was affordable | 6 | 4
  Administered at appointments that I could schedule | 2 | 1
  Administered quickly once arrived at appt | 2 | 3
  Administered at setting that had convenient hours | 3 | 7
  Ensured regular monitoring by healthcare providers | 22 | 10
  Administered by skilled healthcare providers | 24 | 18
  IV antibiotic therapy made me feel better | 19 | 16
  Allowed to receive care for skin infection at home | 7 | 9
  Convenient to administer by self/caregiver at home | 4 | 0
  Other | 3 | 1
  Not satisfied with receiving IV antibiotic therapy | 3 | 2

21. Secondary Outcome: Patient Satisfaction With Care: Factors Contributing to Dissatisfaction With Receiving IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: as for outcome 20
Measure: Number; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 33
Participants
  Got in the way of work/school | 11 | 3
  Got in way of performing daily normal activities | 11 | 3
  Got in the way of providing care to others | 5 | 1
  IV antibiotic therapy was expensive | 2 | 0
  Required me to make appointments | 0 | 0
  Administered at healthcare setting w/limited hours | 0 | 0
  Required traveling to and from appointments | 0 | 1
  Required to wait to be seen by provider | 0 | 5
  IV antibiotic therapy took too long to administer | 4 | 1
  Administered too frequently | 4 | 1
  Required having a PICC or central line inserted | 7 | 2
  Caused an IV site infection | 1 | 0
  IV antibiotic therapy made me feel worse | 10 | 3
  Not adequately monitored by healthcare providers | 3 | 0
  Not administered by skilled healthcare providers | 0 | 0
  IV antibiotic therapy made me feel concerned | 7 | 3
  Required a nurse/healthcare worker coming to home | 0 | 1
  Required administration to self/caregiver at home | 0 | 1
  Other | 1 | 0
  Not dissatisfied w/receiving IV antibiotic therapy | 19 | 22

22. Secondary Outcome: Patient Satisfaction With Care: IV Therapy Hindering Normal Activities of Daily Living
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: FAS Population. 43 & 34 patients provided any survey data in the usual care group & new critical pathway group; 40 & 32 patients completed all survey questions in the usual care group & new critical pathway group; 42 & 33 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 42 | 33
Participants
  None of the time | 17 | 26
  A little of the time | 4 | 5
  Some of the time | 3 | 0
  Most of the time | 6 | 1
  All of the time | 12 | 1

23. Secondary Outcome: Patient Satisfaction With Care: Concerned About Receiving Your IV Therapy
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 42 | 33
Participants
  None of the time | 23 | 26
  A little of the time | 13 | 4
  Some of the time | 3 | 1
  Most of the time | 1 | 1
  All of the time | 2 | 1

24. Secondary Outcome: Patient Satisfaction With Care: Satisfied With the Number of IV Infusions Received Per Day
Description: as for outcome 14
Time Frame: 14 Days
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 33
scores on a scale | 7.3 (2.63) | 8.7 (1.89)

25. Secondary Outcome: Patient Satisfaction With Care: Satisfaction With the Average Time to Administer Each IV
Description: as for outcome 14
Time Frame: 14 Days
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 33
scores on a scale | 7.5 (2.58) | 8.9 (1.9)

26. Secondary Outcome: Patient Satisfaction With Care: Regimen Preferred if Treated Again for a Similar Skin Infection With IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: FAS Population. 43 & 34 patients provided any survey data in the usual care group & new critical pathway group; 40 & 32 patients completed all survey questions in the usual care group & new critical pathway group; 43 & 34 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
Participants
  Regimen 1 | 28 | 33
  Regimen 2 | 6 | 0
  Regimen 3 | 9 | 1

27. Secondary Outcome: Patient Satisfaction With Care: Time Willing to Spend Receiving Each IV
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: FAS Population. 43 & 34 patients provided any survey data in the usual care group & new critical pathway group; 40 & 32 patients completed all survey questions in the usual care group & new critical pathway group; 41 & 34 patients answered this survey question in the usual care group & new critical pathway group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 41 | 34
Participants
  About 30 minutes or less | 23 | 22
  About 1 hour | 10 | 10
  About 1.5 to 2 hours | 5 | 1
  About 3 hours or longer | 3 | 1

28. Secondary Outcome: Patient Satisfaction With Care: Find Value in a Physician
Description: Patient satisfaction with care as assessed through the ABSSSI Patient Satisfaction Survey (patient reported).
Time Frame: 14 Days
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
Participants
  Definitely not | 1 | 1
  Probably not | 1 | 1
  Probably so | 7 | 2
  Definitely so | 34 | 30

29. Secondary Outcome: Patient Work and Productivity Loss as Assessed Through the Work Productivity and Activity Impairment Questionnaire
Time Frame: Day 10-14
Population: FAS population. 43 and 34 patients provided any survey data in the usual care group and the new critical pathway group, respectively.14 and 9 patients completed all survey questions in the usual care group and new critical pathway group, respectively. 17 and 20 patients were employed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 43 | 34
Percentage
  Absenteeism: number analyzed (Participants) | 17 | 16
  Absenteeism | 49.9 (38.49) | 36.7 (46.09)
  Impairment while working: number analyzed (Participants) | 14 | 9
  Impairment while working | 47.9 (40.03) | 8.9 (9.28)
  Overall work impairment: number analyzed (Participants) | 14 | 9
  Overall work impairment | 59.3 (39.16) | 18.0 (23.39)
  Activity impairment: number analyzed (Participants) | 42 | 33
  Activity impairment | 60.2 (38.85) | 18.5 (26.23)

30. Secondary Outcome: Patient Health-related Quality of Life (HRQoL) Assessed by the Short Form 12 (SF-12) 12-Item Patient Questionnaire
Description: The SF-12 yields a physical and a mental health component summary score (referred to as physical component summary score [PCS] and mental component summary score [MCS]). The PCS and MCS follow a t-score distribution, i.e. mean of 50 and standard deviation of 10 in the general US population, meaning all scores above or below 50 are above and below the average, respectively, in the US general population.
Time Frame: Day 14
Population: FAS population. 43 and 34 patients provided any survey data in the usual care group and the new critical pathway group, respectively. 42 and 34 patients completed all survey questions in the usual care group and new critical pathway group, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 42 | 34
score on a scale
  Mental Health Component Score | 43.9 (10.28) | 50.8 (10.85)
  Physical Health Component Score | 40.5 (11.37) | 46.3 (11.15)

31. Secondary Outcome: Healthcare Costs
Description: Cost of hospital inpatient stays, ED visits, healthcare visits, procedures, and biological tests
Time Frame: 44 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Usual Care | New Critical Pathway
Number analyzed (Participants) | 48 | 42
USD | 13772.9 (7166.95) | 9421.6 (7122.57)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 44 days. Initial care is the date of enrollment to 10-14 days and follow-up is 30 days after initial care.
Arm/Group | Usual Care | New Critical Pathway
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/48 | 3/42
Other Adverse Events (participants affected / at risk) | 0/48 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=48) | New Critical Pathway (N=42)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=48) | New Critical Pathway (N=42)
Pyrexia (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03233438/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT03233438/SAP_001.pdf